CLINICAL TRIAL: NCT01207388
Title: A Confirmatory Multicenter, Single-arm Study to Assess the Efficacy, Safety, and Tolerability of the BiTE® Antibody Blinatumomab in Adult Patients With Minimal Residual Disease (MRD) of B-precursor Acute Lymphoblastic Leukemia (BLAST)
Brief Title: Confirmatory Phase II Study of Blinatumomab (MT103) in Patients With Minimal Residual Disease of B-precursor Acute Lymphoblastic Leukemia (ALL)
Acronym: BLAST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen Research (Munich) GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT103-203
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: Blinatumomab; MRD; B-ALL; Minimal residual disease; adult ALL; Leukemia; ALL; Lymphatic diseases; Lymphoproliferative disorders; bispecific antibody; anti-CD19; Immunotherapeutic treatment
MeSH Terms: conditions — Burkitt Lymphoma; Neoplasm, Residual; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Lymphatic Diseases; Lymphoproliferative Disorders | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Blinatumomab (Experimental): Participants received blinatumomab as a continuous intravenous infusion at a constant flow rate of 15 μg/m²/day over 28 days followed by an infusion-free period of 14 days for up to 4 cycles of treatment.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Continuous intravenous infusion
  Other Names: AMG 103; MT103; BLINCYTO™

SUMMARY:
The purpose of this study is to confirm whether the bispecific T cell engager blinatumomab (MT103) is effective, safe and tolerable in the treatment of ALL patients with minimal residual disease.

DETAILED DESCRIPTION:
The detection of minimal residual disease (MRD) after induction therapy and/or consolidation therapy is an independent prognostic factor for poor outcome of adult ALL. No standard treatments are available for patients with MRD-positive B-precursor ALL. Blinatumomab (MT103) is a bispecific single-chain antibody construct designed to link B cells and T cells resulting in T-cell activation and a cytotoxic T-cell response against cluster of differentiation (CD)19 expressing cells. The purpose of this study is to confirm whether the bispecific T-cell engager blinatumomab (MT103) is effective, safe and tolerable in the treatment of ALL patients with minimal residual disease.

Participants will receive up to four 4-week cycles of intravenous blinatumomab treatment followed by an infusion-free period of 14 days. A safety follow-up will be performed 30 days after the end of the last infusion and efficacy follow-ups will occur until 24 months after treatment start. Participants will be followed for up to 5 years after the start of treatment for survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with B-precursor ALL in complete hematological remission after at least 3 intense chemotherapy blocks
* Presence of minimal residual disease at a level of ≥ 10^-3
* Availability of bone marrow specimen from primary diagnosis for clone-specific MRD assessment
* Negative human immunodeficiency virus (HIV) test, negative hepatitis B (HbsAg) test and hepatitis C virus (anti-HCV) test
* Negative pregnancy test in women of childbearing potential
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

* Presence of circulating blasts or current extra-medullary involvement by ALL
* History of relevant central nervous system (CNS) pathology or current CNS pathology
* Prior allogeneic hematopoietic stem cell transplant (HSCT)
* Eligibility for treatment with tyrosine-kinase inhibitors (TKI)
* Systemic cancer chemotherapy within 2 weeks prior to study treatment
* Therapy with monoclonal antibodies (rituximab, alemtuzumab) within 4 weeks prior to study treatment
* Previous treatment with blinatumomab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2010-11; Primary Completion 2014-02 (Actual); Study Completion 2019-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Bargou, MD, Principal Investigator — Medizinische Klinik und Poliklinik II, Würzburg; Nicola Gökbuget, MD, Principal Investigator — Klinikum der Goethe Universität Frankfurt
Locations (75):
- Austria (4):
  - 1102 - LKH Graz, Graz
  - 1107 - Krankenhaus der Elisabethinen, Linz
  - 1106, Salzburg
  - 1101 - AKH Wien, Vienna
- Belgium (5):
  - 1504, Antwerp
  - 1505, Bruges
  - 1502 - Cliniques Universitaires de Saint-Luc, Brussels
  - 1503, Ghent
  - 1501 - Cliniques Universitaires UCL de Mont Godinne, Yvoir
- France (10):
  - 1211 - CHU d'Angers, Angers
  - 1210 - CHU de Besançon, Besançon
  - 1206 - Hôpital de Pontoise, Cergy-Pontoise
  - 1205 - CHU Henri Mondor, Créteil
  - 1209 - CHU de Lyon, Lyon
  - 1212 - Hôpital de l'hôtel Dieu, Nantes
  - 1213 - Centre Hospitalier Universitaire de Nice, Nice
  - 1201 - Hôpital Saint Louis, Paris
  - 1202 - CHU de Bordeaux - Hôpital Haut Lévêque, Pessac
  - 1208 - CHU de Purpan, Toulouse
- Germany (17):
  - 1011 - Charité Berlin, Berlin
  - 1022 - Universitätsklinkum Carl Gustav Carus Dresden, Dresden
  - 1009 - Universitätsklinikum Essen, Essen
  - 1002 - Klinikum der Goethe Universität, Frankfurt
  - 1014 - Asklepiosklinik St. Georg, Hamburg
  - 1018 - Medizinische Hochschule Hannover, Hanover
  - 1012 - Universitätsklinikum Heidelberg, Heidelberg
  - 1003 - Universitätsklinikum Schleswig-Holstein, Kiel
  - 1019 - Universitätsklinikum Leipzig, Leipzig
  - 1010 - Klinikum der Universität München - Großhadern, Munich
  - 1004 - Universitätsklinikum Münster, Münster
  - 1016 - Universitätsklinikum Regensburg, Regensburg
  - 1020 - Universitätsklinikum Rostock, Rostock
  - 1007 - Robert-Bosch-Krankenhaus, Stuttgart
  - 1015 - Universitätsklinikum Tübingen, Tübingen
  - 1005 - Universitätsklinikum Ulm, Ulm
  - 1001 - Julius-Maximilians-Universität Würzburg, Würzburg
- Italy (12):
  - 1301 - Ospedali Riuniti di Bergamo, Bergamo
  - 1303 - Istituto di Ematologia "L.& A.Seràgnoli" Azienda, Bologna
  - 1314 - Azienda Ospedaliera Spedali Civili Brescia, Brescia
  - 1313 - Universita di Catania, Catania
  - 1312 - Azienda Ospedaliera Universitaria San Martino, Genoa
  - 1305 - Ospedale San Gerardo, Monza
  - 1309 - Azienda Ospedaliera Antonio Cardarelli, Napoli
  - 1308 - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - 1302 - Università La Sapienza di Roma, Rome
  - 1310 - Fondazione Policlinico Tor Vergata, Rome
  - 1315 - Azienda Ospedaliero-Universitaria S. Giovanni Battista (Le Molinette), Torino
  - 1311 - Azienda Ospedaliera di Verona, Verona
- Netherlands (2):
  - 2204 - UMC Groningen, Groningen
  - 2201 - Daniel Den Hoed Hospitaal, Rotterdam
- Poland (7):
  - 1905 - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok
  - 1907 - Uniwersyteckie Centrum Kliniczne, Gdansk
  - 1908 - Swietokrzyskie Centrum Onkologii, Kielce
  - 1902 - Uniwersytet Medyczny w Lublinie, Lublin
  - 1901 - Klinika Hematologii - Instytut Hematologii i Transfuzjologii, Warsaw
  - 1906 - MTZ Clinical Research Sp. z o.o., Warsaw
  - 1904 - Samodzielny Publiczny, Wroclaw
- Romania (4):
  - 2101 - Institutul Clinic Fundeni, Hematologie II, Bucharest
  - 2102 - Spitalul Clinic Coltea, Hematologie, Bucharest
  - 2106 - Institutul Oncologic "Prof. Dr. I. Chiricuta", Cluj-Napoca
  - 2105 - Institutul Regional de Oncologie, Iași
- Russia (2):
  - 2001 - Russian Hematology Research Center, Moscow
  - 2003 - Municipal Hospital No. 15, Saint Petersburg
- Spain (7):
  - 1402 - Complexo Hospitalario Universitario A Coruña, A Coruña
  - 1401 - ICO Hospital Germans Trias I Pujol, Badalona
  - 1404 - Hospital Clínic Servei d´Hematologia, Barcelona
  - 1408 - Hospital 12 de Octubre, Madrid
  - 1405 - Hospital Universitari Son Espases, Mallorca
  - 1407 - Unidad de Citogenética Oncológica, Salamanca
  - 1406 - Hospital Universitari i Politècnic La Fe de Valencia, Valencia
- United Kingdom (5):
  - 1605 - Queen Elizabeth Hospital, Birmingham
  - 1602 - Bristol Royal Infirmary, Bristol
  - 1604 - University Hospital of Wales, Cardiff
  - 1601 - Royal Free Hospital, London
  - 1607 - Nottingham City Hospital NHS Trust, Nottingham

REFERENCES:
- [Derived] Chevallier P. Should patients with Ph-negative acute lymphoblastic leukaemia who reach minimal residual disease negativity have HSCT? Lancet Haematol. 2024 Jan;11(1):e12-e13. doi: 10.1016/S2352-3026(23)00365-4. No abstract available. PMID 38135369
- [Derived] Gokbuget N, Zugmaier G, Dombret H, Stein A, Bonifacio M, Graux C, Faul C, Bruggemann M, Taylor K, Mergen N, Reichle A, Horst HA, Havelange V, Topp MS, Bargou RC. Curative outcomes following blinatumomab in adults with minimal residual disease B-cell precursor acute lymphoblastic leukemia. Leuk Lymphoma. 2020 Nov;61(11):2665-2673. doi: 10.1080/10428194.2020.1780583. Epub 2020 Jul 3. PMID 32619115
- [Derived] Jen EY, Xu Q, Schetter A, Przepiorka D, Shen YL, Roscoe D, Sridhara R, Deisseroth A, Philip R, Farrell AT, Pazdur R. FDA Approval: Blinatumomab for Patients with B-cell Precursor Acute Lymphoblastic Leukemia in Morphologic Remission with Minimal Residual Disease. Clin Cancer Res. 2019 Jan 15;25(2):473-477. doi: 10.1158/1078-0432.CCR-18-2337. Epub 2018 Sep 25. PMID 30254079
- [Derived] Gokbuget N, Dombret H, Bonifacio M, Reichle A, Graux C, Faul C, Diedrich H, Topp MS, Bruggemann M, Horst HA, Havelange V, Stieglmaier J, Wessels H, Haddad V, Benjamin JE, Zugmaier G, Nagorsen D, Bargou RC. Blinatumomab for minimal residual disease in adults with B-cell precursor acute lymphoblastic leukemia. Blood. 2018 Apr 5;131(14):1522-1531. doi: 10.1182/blood-2017-08-798322. Epub 2018 Jan 22. PMID 29358182
- [Derived] Zhu M, Wu B, Brandl C, Johnson J, Wolf A, Chow A, Doshi S. Blinatumomab, a Bispecific T-cell Engager (BiTE((R))) for CD-19 Targeted Cancer Immunotherapy: Clinical Pharmacology and Its Implications. Clin Pharmacokinet. 2016 Oct;55(10):1271-1288. doi: 10.1007/s40262-016-0405-4. PMID 27209293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was open to adults with a diagnosis of minimal residual disease (MRD; ≥ 10-³ leukemic cells) -positive B-precursor acute lymphoblastic leukemia (ALL) who were in complete hematologic remission.
Groups:
- Blinatumomab: Participants received blinatumomab as a continuous intravenous infusion at a constant flow rate of 15 μg/m²/day over 28 days followed by an infusion-free period of 14 days for up to 4 cycles of treatment.
  Participants suitable for allogeneic hematopoietic stem cell transplant (HSCT) after treatment with at least 1 cycle of blinatumomab may have undergone allogeneic HSCT instead of receiving further cycles with blinatumomab.
Period: Overall Study
Arm/Group | Blinatumomab
Started | 116
Completed | 48
Not Completed | 68
Not completed — Death | 67
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (all participants who received any infusion of blinatumomab)
Arm/Group | Blinatumomab
Number analyzed (Participants) | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (16.4)
Age, Customized [Number; unit: participants]
  ≥ 18 and <35 years | 36
  ≥ 35 and < 55 years | 41
  ≥ 55 and < 65 years | 24
  ≥ 65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 68
Race/Ethnicity, Customized [Number; unit: participants] — Race was not permitted to be collected in France.
  participants
    White | 102
    Asian | 1
    Mixed | 1
    Unknown | 12
Philadelphia Chromosome Disease Status [Number; unit: participants]
  Positive | 5
  Negative | 111
Confirmed t(4;11) Translocation / MLL-AF4+ ALL [Count of Participants; unit: Participants] — t(4;11)(q21;q23) translocation, resulting in the fusion of the mixed lineage leukemia (MLL) gene on chromosome 11 and the AF4 gene on chromosome 4
  Participants
    Yes | 5
    No | 88
    Unknown | 23
MRD Level at Baseline by Central Laboratory [Number; unit: participants] — Measured by polymerase chain reaction (PCR) performed on bone marrow and assessed by the central laboratory; Lower limit of quantification was at least 10^-4 leukemic cells.
  participants
    ≥ 10^-1 and < 1 | 9
    ≥ 10^-2 and < 10^-1 | 45
    ≥ 10^-3 and < 10^-2 | 52
    < 10^-3 | 3
    Below Lower Limit of Quantification | 5
    Unknown | 2
White Blood Cells at First Diagnosis [Number; unit: participants]
  ≤ 30,000/mL | 78
  > 30,000/mL | 18
  Unknown | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Minimal Residual Disease (MRD) Response Within the First Treatment Cycle
Description: At the end of the first treatment cycle (Day 29) a bone marrow aspiration/biopsy was performed and evaluated by the central MRD laboratory.
  Complete MRD response is defined as no polymerase chain reaction (PCR) amplification of individual rearrangements of immunoglobulin (Ig)- or T-cell receptor (TCR)-genes detected after completion of the first cycle.
Time Frame: During the first cycle (6 weeks)
Population: Primary endpoint full analysis set (Prim EP FAS) included all participants with an Ig TCR PCR MRD assay with the minimum required sensitivity of 1 x 10^-4 at central lab established at Baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 113
percentage of participants | 77.0 [68.1 to 84.4]

2. Secondary Outcome: Hematological Relapse-free Survival (RFS)
Description: Hematological RFS was measured from first dose of blinatumomab until the first assessment of documented relapse (either hematological or extramedullary), secondary leukemia, or death due to any cause. Participants without a documented relapse, or death due to any cause were censored at the time of their last hematological assessment. Participants who received chemotherapy for relapsed or persistent MRD or for any other reason after treatment with blinatumomab, or HSCT after treatment with blinatumomab, before hematological or extramedullary relapse, or death occurred were censored at the start of chemotherapy or HSCT, respectively.
  Hematological relapse was defined as unequivocal detection of > 5% leukemia cells in bone marrow as measured by cytological, microscopic assessment, presence of circulating leukemia blasts, or extramedullary leukemia (whichever occurred first).
  The 18-month Kaplan-Meier estimate of hematological RFS is reported.
Time Frame: 18 months, up to the data cut-off date of 05 August 2015
Population: Full analysis set participants who were in hematological complete remission at treatment start, excluding Philadelphia-positive participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 110
percentage of participants | 54 [33 to 70]

3. Secondary Outcome: Overall Survival
Description: Overall survival was measured from the first treatment with blinatumomab until death due to any cause. Participants who did not die were censored at their last contact date.
Time Frame: Until the data cut-off date of 05 August 2015; median time on study was 18.3 months.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 116
months | 36.5 [19.2 to NA] — Not estimable at the time of analysis due to the low number of events

4. Secondary Outcome: 100-Day Mortality After Allogeneic Hematopoietic Stem Cell Transplant
Description: The mortality rate within 100 days after allogeneic HSCT was defined as the Kaplan-Meier estimate of the percentage of participants dying within 100 days after the day of the first allogeneic HSCT.
Time Frame: 100 days after HSCT, as of the data cut-off date of 05 August 2015
Population: Full analysis set participants who underwent HSCT prior to relapse (hematological or extramedullary) excluding Philadelphia-positive participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 74
percentage of participants | 7 [3 to 15]

5. Secondary Outcome: Time to Hematological Relapse
Description: Time to hematological relapse was measured from the start of treatment with blinatumomab until hematological or extramedullary relapse. Participants who died or received HSCT or post-blinatumomab chemotherapy after treatment with blinatumomab were censored at their last hematological assessment prior to death or HSCT or post-blinatumomab chemotherapy (whichever occurred first).
Time Frame: Until the data cut-off date of 05 August 2015; median time on study was 18.3 months.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 110
months | NA [7.1 to NA] — Data not estimable due to the low number of events

6. Secondary Outcome: Duration of Complete MRD Response
Description: The duration of MRD response was analyzed as the time from onset of MRD negativity until MRD or hematological relapse or date of last confirmation of negative MRD status. Participants who received chemotherapy or HSCT after treatment with blinatumomab, before hematological or extramedullary relapse were censored at the start of chemotherapy or HSCT, respectively.
  MRD relapse is defined as the reappearance of individual rearrangements of Ig- or TCR-genes ≥ lower limit of quantification (LLOQ) for at least 1 individual marker measured by an assay with a sensitivity of minimum 10^-4. Hematological relapse is defined as the unequivocal detection of > 5% leukemia cells in bone marrow as measured by cytological or microscopic assessment, presence of circulating leukemia blasts, or extramedullary leukemia.
Time Frame: Until the data cut-off date of 05 August 2015; median time on study was 18.3 months.
Population: Full analysis set participants who were in hematological complete remission at treatment start, excluding Philadelphia-positive participants, who had an MRD complete response at cycle 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 85
months | 45.0 [6.5 to 45.0]

7. Secondary Outcome: Change in MRD Level From Baseline to End of Cycle 1 in Non-MRD Responders
Description: MRD level was measured by polymerase chain reaction (PCR) performed on bone marrow and assessed by the central laboratory. An MRD level of 10^-n corresponds to residual leukemia cells at a frequency of 1 per 10ⁿ bone marrow cells.
Time Frame: Baseline and end of cycle 1 (6 weeks)
Population: Full analysis set participants who were in hematological complete remission at treatment start, with no MRD Response in the first treatment cycle, excluding Philadelphia-positive participants.
Measure: Count of Participants; unit: Participants
Groups:
- Cycle 1 MRD 10^-5: Participants with an MRD level 10^-5 at the end of cycle 1.
- Cycle 1 MRD 10^-4: Participants with an MRD level 10^-4 at the end of cycle 1.
- Cycle 1 MRD 10^-3: Participants with an MRD level 10^-3 at the end of cycle 1.
- Cycle 1 MRD 10^-2: Participants with an MRD level 10^-2 at the end of cycle 1.
- Cycle 1 MRD 10^-1: Participants with an MRD level 10^-1 at the end of cycle 1.
- Cycle 1 MRD Unknown: Participants with an unknown MRD level at the end of cycle 1.
Arm/Group | Cycle 1 MRD 10^-5 | Cycle 1 MRD 10^-4 | Cycle 1 MRD 10^-3 | Cycle 1 MRD 10^-2 | Cycle 1 MRD 10^-1 | Cycle 1 MRD Unknown
Number analyzed (Participants) | 2 | 13 | 4 | 0 | 2 | 2
Participants
  Baseline MRD Unknown | 0 | 1 | 0 |  | 0 | 0
  Baseline MRD 10^-5 | 0 | 0 | 0 |  | 0 | 0
  Baseline MRD 10^-4 | 0 | 1 | 0 |  | 0 | 0
  Baseline MRD 10^-3 | 1 | 6 | 2 |  | 1 | 0
  Baseline MRD 10^-2 | 0 | 5 | 2 |  | 1 | 0
  Baseline MRD 10^-1 | 1 | 0 | 0 |  | 0 | 2

8. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) were evaluated for severity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4, as follows:
  Grade 1 - Mild AE;
  Grade 2 - Moderate AE;
  Grade 3 - Severe AE;
  Grade 4 - Life-threatening or disabling AE;
  Grade 5 - Death.
  The investigator used medical judgment to determine if there was a causal relationship (ie, related, unrelated) between an adverse event and blinatumomab.
  An AE was considered "serious" if it resulted in death, was life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant incapacity or substantial disruption to conduct normal life functions, was a congenital anomaly or birth defect or was a medically important condition.
Time Frame: From the first dose of blinatumomab until 30 days after last dose; the median treatment duration was 55 days.
Population: All participants who received any infusion of blinatumomab.
Measure: Number; unit: participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 116
participants
  Any adverse event | 116
  Serious adverse events | 73
  Adverse events ≥ CTC grade 3 | 71
  Adverse events ≥ CTC grade 4 | 33
  Fatal adverse events | 2
  AEs leading to discontinuation of blinatumomab | 20
  AEs leading to interruption of blinatumomab | 36
  Treatment-related adverse events | 112
  Treatment-related serious adverse events | 60
  Treatment-related adverse events ≥ CTC grade 3 | 60
  Treatment-related adverse events ≥ CTC grade 4 | 26
  Treatment-related fatal adverse events | 1

9. Secondary Outcome: Change From Baseline in EORTC-QLQ-C30 Scales
Description: The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Insomnia, Appetite Loss, Constipation, Diarrhea, Financial Impact).
  For each of these scales, scores range from 0 to 100. For the GHS and 5 functional scales a high score indicates better global health status/functioning and a positive change from baseline indicates improvement. For the 9 symptom scales, a high score indicates a higher level of symptoms, and a negative change from Baseline indicates an improvement in symptoms.
  The maximum changes from baseline to cycles 1 through 4 and the change from baseline to the end of the core study are reported.
Time Frame: Baseline and the end of each treatment cycle (day 29 of each cycle) and 30 days after end of the last infusion (end of the core study, a maximum of 26 weeks).
Population: FAS with available data at relevant time points. For maximum change, the change from baseline was calculated using subset of FAS with available data (baseline and post-baseline) at the end of each cycle. The number analyzed are the number of subjects with available data at the time point at which maximum change from baseline was observed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Maximum Change From Baseline in Cycles 1 - 4 | Change From Baseline at End of Core Study
Number analyzed (Participants) | 111 | 74
units on a scale
  Global Health Status: number analyzed (Participants) | 26 | 74
  Global Health Status | 9.0 (4.2) | 3.9 (2.4)
  Physical Functioning: number analyzed (Participants) | 26 | 74
  Physical Functioning | 2.6 (2.3) | 2.2 (1.9)
  Role Functioning: number analyzed (Participants) | 15 | 72
  Role Functioning | 12.2 (8.5) | 1.4 (3.5)
  Emotional Functioning: number analyzed (Participants) | 26 | 74
  Emotional Functioning | 6.5 (4.9) | 5.3 (2.7)
  Cognitive Functioning: number analyzed (Participants) | 15 | 74
  Cognitive Functioning | -3.3 (5.2) | -2.3 (2.5)
  Social Functioning: number analyzed (Participants) | 15 | 74
  Social Functioning | 12.2 (8.5) | 14.9 (3.8)
  Fatigue Symptom: number analyzed (Participants) | 15 | 74
  Fatigue Symptom | -5.9 (5.5) | -5.4 (2.4)
  Nausea and Vomiting Symptom: number analyzed (Participants) | 26 | 73
  Nausea and Vomiting Symptom | -4.5 (4.7) | -2.3 (2.0)
  Pain Symptom: number analyzed (Participants) | 26 | 74
  Pain Symptom | 3.8 (3.6) | -1.4 (2.7)
  Dyspnea Symptom: number analyzed (Participants) | 26 | 74
  Dyspnea Symptom | -9.0 (4.7) | -0.9 (2.9)
  Insomnia Symptom: number analyzed (Participants) | 26 | 73
  Insomnia Symptom | -2.6 (3.2) | 3.7 (3.5)
  Appetite Loss Symptom: number analyzed (Participants) | 15 | 73
  Appetite Loss Symptom | -17.8 (6.4) | -9.1 (3.4)
  Constipation Symptom: number analyzed (Participants) | 26 | 74
  Constipation Symptom | -5.1 (3.6) | 0.0 (2.2)
  Diarrhea Symptom: number analyzed (Participants) | 26 | 74
  Diarrhea Symptom | 5.1 (5.5) | 0.0 (2.3)
  Financial Difficulties Symptom: number analyzed (Participants) | 26 | 72
  Financial Difficulties Symptom | -5.1 (4.8) | -0.9 (2.9)

10. Secondary Outcome: Change From Baseline in EuroQoL 5-Dimension (EQ-5D) Scales
Description: The EQ-5D is a self-administered questionnaire which captures 3 basic types of information: a descriptive profile (health state index) and the overall health rating using a visual analog scale. The health state index measures mobility, self-care, usual activities, pain/discomfort and anxiety/depression on scales from no problems (score = 1), some problems (score = 2), to extreme problems (score = 3). For each dimension the mean change from baseline was calculated at the end of each treatment cycle and at the end of the core study. The maximum observed change from baseline during cycles 1 to 4 and the change from baseline at the end of the core study are reported for each dimension.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Maximum Change From Baseline in Cycles 1 - 4 | Change From Baseline at End of Core Study
Number analyzed (Participants) | 112 | 75
units on a scale
  Mobility: number analyzed (Participants) | 14 | 75
  Mobility | -0.2 (0.1) | 0.0 (0.1)
  Self-care: number analyzed (Participants) | 13 | 73
  Self-care | -0.1 (0.1) | 0.0 (0.0)
  Usual Activities: number analyzed (Participants) | 27 | 75
  Usual Activities | -0.1 (0.1) | -0.1 (0.1)
  Pain/Discomfort: number analyzed (Participants) | 14 | 75
  Pain/Discomfort | -0.2 (0.2) | -0.1 (0.1)
  Anxiety/Depression: number analyzed (Participants) | 56 | 75
  Anxiety/Depression | -0.2 (0.1) | -0.1 (0.1)

11. Secondary Outcome: Resource Utilization: Number of Participants Reporting Use of Transfusion of Blood Products
Time Frame: From first dose of study drug through the end of follow-up; median (minimum, maximum) time on study was 33.8 (1, 62) months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 116
Participants
  Overall | 14
  Cycle 1 | 5
  Cycle 2 | 8
  Cycle 3 | 0
  Cycle 4 | 1
  Follow-up period | 0

12. Secondary Outcome: Resource Utilization: Duration of Hospitalization
Time Frame: as for outcome 11
Population: Full analysis set
Measure: Median (Full Range); unit: days
Arm/Group | Blinatumomab
Number analyzed (Participants) | 116
days | 14.0 [3 to 63]

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment until the end of the follow-up period; median (minimum, maximum) time on study was 33.8 (1, 62) months. Adverse events are reported from the first dose of blinatumomab until 30 days after last dose; the median treatment duration was 55 days.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Blinatumomab
All-Cause Mortality (participants affected / at risk) | 67/116
Serious Adverse Events (participants affected / at risk) | 73/116
Other Adverse Events (participants affected / at risk) | 111/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab (N=116)
Anaemia (Blood and lymphatic system disorders) | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Device issue (General disorders) | 1
Device malfunction (General disorders) | 2
Fatigue (General disorders) | 1
Gait disturbance (General disorders) | 1
Infusion site extravasation (General disorders) | 1
Product contamination microbial (General disorders) | 1
Puncture site pain (General disorders) | 1
Pyrexia (General disorders) | 17
Thrombosis in device (General disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Cytokine release syndrome (Immune system disorders) | 2
Hypersensitivity (Immune system disorders) | 2
Acinetobacter bacteraemia (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Cystitis klebsiella (Infections and infestations) | 1
Device related infection (Infections and infestations) | 3
H1N1 influenza (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Staphylococcal infection (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection staphylococcal (Infections and infestations) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 5
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Body temperature increased (Investigations) | 1
C-reactive protein increased (Investigations) | 4
Hepatic enzyme increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Prothrombin time prolonged (Investigations) | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 6
Ataxia (Nervous system disorders) | 2
Cognitive disorder (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 6
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Intention tremor (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Motor dysfunction (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 8
Agitation (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab (N=116)
Anaemia (Blood and lymphatic system disorders) | 6
Leukopenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 14
Constipation (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 22
Nausea (Gastrointestinal disorders) | 27
Vomiting (Gastrointestinal disorders) | 26
Chills (General disorders) | 30
Fatigue (General disorders) | 27
Pyrexia (General disorders) | 99
Device related infection (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 8
Blood immunoglobulin G decreased (Investigations) | 6
C-reactive protein increased (Investigations) | 6
Weight increased (Investigations) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 18
Hypomagnesaemia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 15
Back pain (Musculoskeletal and connective tissue disorders) | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Aphasia (Nervous system disorders) | 9
Dizziness (Nervous system disorders) | 9
Headache (Nervous system disorders) | 44
Paraesthesia (Nervous system disorders) | 6
Tremor (Nervous system disorders) | 28
Insomnia (Psychiatric disorders) | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Night sweats (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 11
Hypertension (Vascular disorders) | 7
Hypotension (Vascular disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.